CLINICAL TRIAL: NCT02960321
Title: Myocardial Injury Related to Coronary Angiography in the Era of High-sensitivity Cardiac Troponin I
Brief Title: Troponin Release Induced by Procedure - Czech
Acronym: TRIP-CZ
Status: Completed | Type: Observational
Sponsor: Tomas Bata Hospital, Czech Republic (Other)
Responsible Party: Sponsor
Other Study IDs: BN112016
Record Dates: First submitted 2016-11-06; First posted 2016-11-09 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Coronary Artery Disease
Keywords: myocardial injury; high-sensitivity troponin I; periprocedural myocardial infarction
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CAG without PCI: Diagnostic coronary angiography only
- CAG with PCI: Diagnostic coronary angiography and subsequent percutaneous coronary intervention (PCI)

SUMMARY:
A prospective study aiming to analyse the relation between different variables and high sensitivity troponin I (hsTnI) elevation within a group of patients undergoing a coronary angiography with or without subsequent percutaneous coronary intervention.

DETAILED DESCRIPTION:
The study tries to seek potential causes and context of subclinical myocardial injury within patients with baseline concentration of hsTnI below the 99th percentile value upper reference limit or with demonstrated fall of hsTnI levels.

ELIGIBILITY:
Inclusion Criteria:

* stable or unknown coronary artery disease
* acute coronary syndrome without ST-segment elevation meeting the criteria of low risk with demonstrated fall of cTn levels

Exclusion Criteria:

* acute coronary syndrome with persistent ST-segment elevation
* acute coronary syndrome without ST-segment elevation meeting the criteria of high or intermediate risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients referred for coronary angiography (CAG): stable patients with presumed coronary artery disease, or those referred for acute coronary syndrome without ST-segment elevation (NSTE-ACS) meeting the criteria of low risk with demostrated fall of cTn levels, or patients prepared for cardiac surgery.
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2016-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Subclinical myocardial injury | up to 24 hours after procedure

SECONDARY OUTCOMES:
Postprocedural myocardial infarction | up to 24 hours after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Martin Griva, MD, Principal Investigator — Cardiac Center for Adults, Tomas Bata Hospital, Zlin, Czech Republic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Griva M, Stastny J, Kopriva P, Slabak M, Coufal Z, Jarkovsky J, Svoboda M, Salek T, Sukupova L, Taborsky M. Selective coronary angiography, percutaneous coronary intervention and asymptomatic peri-procedural myocardial injury. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2019 Dec;163(4):324-330. doi: 10.5507/bp.2018.066. Epub 2018 Nov 6. PMID 30398220